CLINICAL TRIAL: NCT06657573
Title: AI-enabled Vaccine Chatbot for Improving Influenza Vaccination Uptake in Children: a Cluster Randomized Trial
Brief Title: Vaccine Chatbot for Improving Influenza Vaccination Uptake
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhiyuan Hou, Associate professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Fudan Univeristy
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Influenza Vaccines
Keywords: Influenza vaccine; vaccination; vaccine confidence; AI; Chatbot
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Influenza Vaccine Chatbot Intervention group (Experimental): In this arm, participants will receive a vaccine chatbot intervention for one and a half months. The AI-enabled influenza vaccine chatbot can be accessed online through WeChat or any web browsers, where people can ask any questions related to the influenza vaccine and get previously validated answers from the chatbot immediately. The chatbot is available for use at their convenience during the 1.5-month intervention, with invitations sent every ten days to reinforce the engagement.
  Interventions: Behavioral: An AI-enabled chatbot tailored for influenza vaccine consultation
- Control group (No Intervention): The control group will not use the chatbot during the intervention duration.

INTERVENTIONS:
Behavioral: An AI-enabled chatbot tailored for influenza vaccine consultation — The AI-enabled influenza vaccine chatbot can be accessed online through WeChat or any web browsers. The foundation of this chatbot is an expansive knowledge database, constructed with information sourced exclusively from healthcare authorities such as China CDCs and Health Departments, and thoroughly verified by public health experts. This database integrates data on the disease's burden, susceptibility, and severity, along with in-depth details about the vaccines, including their importance, efficacy, safety, and recommended demographics and timing for vaccination. It also covers types and costs of vaccines, societal norms such as vaccination guidelines, expert recommendations, and vaccination trends both in China and internationally. It also includes misinformation and fact-checking contents and provides information about vaccination services such as locations and appointment scheduling.
  Arms: Influenza Vaccine Chatbot Intervention group

SUMMARY:
This study aims to assess the impact of a vaccine chatbot on improving influenza vaccination uptake among children aged between 6 and 59 months through a cluster randomized trial. Specifically, the main questions it seeks to answer are whether an AI-enabled vaccine chatbot will increase the uptake of influenza vaccine among children and their family members, and how it will influence parents' literacy and confidence towards influenza vaccine. It will explore the potential role of vaccine chatbot on vaccination services.

A cluster randomization will be used to assign children to the intervention and control groups. Parents of children in the intervention group will be invited to use the influenza vaccine chatbot online through WeChat, the mostly widely used social media platform in mainland China, or any web browsers. They can ask any questions related to the influenza vaccine and receive validated answers from the chatbot immediately. The intervention will last one and a half months, with invitations sent every ten days to reinforce the engagement. The control group will not use the chatbot during the intervention duration. After the intervention, the uptake, literacy, and confidence towards influenza vaccine will be compared between the intervention and control groups to evaluate the impact of vaccine chatbot.

DETAILED DESCRIPTION:
This is a cluster randomized trial (CRTs) consisting of two arms to evaluate the effectiveness of an AI-enabled vaccine chatbot on influenza vaccination uptake among children aged between 6 and 59 months. Participants regularly visit primary care clinics when they are invited to participate in this trial, and with clinic-days as clusters, a cluster randomization will be used to assign clinic days to the intervention and control groups.

The sample size is calculated based on the primary outcome - the influenza vaccination uptake among children, and the main analysis method, which involves the comparison of differences in vaccination rates between the intervention and control groups after the intervention. According to the vaccination data of study sites, the uptake of influenza vaccine among children aged 6-59 months is around 20% in the previous flu season. In China, influenza vaccination starts in September, and has been available for two months before this trial. Therefore, we assume that the baseline vaccination rate is 10% without the intervention during this trial, and the chatbot intervention would raise this rate by 6 percentage points to 16% at least. We assume a cluster size of 15 children per day per clinic based on routine visiting data. To have 80% power to detect a difference between the group proportions of 0.06, it requires 35 clusters and 525 participants per arm, assuming an intracluster correlation coefficient of 0.005 and a two-sided test with the 0.05 significance level. Assuming at least 10% loss to follow-up, the sample size is 600 participants per arm and 1,200 in total.

Multi-stage sampling will be utilized. Firstly, three representative regions (an urban district, a suburban district, and a rural county) will be selected to represent different economic development levels in China. In each region, four clinics will be selected based on geographical location, economic development, and patient volume. In each clinic, the 6-8 working days will be chosen to conduct this trial, resulting in 72-96 clinic-days (clusters) in 12 clinics in total. In these selected clinic-days, children and their parents regularly visit primary care clinics. All eligible children presenting in the selected clinic-days will be invited to participate by medical staff, and one of their parents will be included in this trial.

Stratified cluster randomized grouping will be employed. All clinic-days will be randomly allocated into intervention group or control group at a 1:1 ratio, stratified by region and clinic, resulting with 36-48 clinic-days per arm. Approximately 400 participants (200 in intervention group; 200 in control group) are expected to participate in this trial in each region, with a total sample size of 1,200 participants, meeting the sample size requirement.

The intervention group will engage with influenza vaccine chatbot for one and a half months, while the control group will receive the standard of care according to the local context, without additional intervention. On the day of the visit, the intervention group will be invited to use the influenza vaccine chatbot online through WeChat or any web browsers, where they can ask any questions related to the influenza vaccine and get validated answers from the chatbot immediately. Staff will be on site to help them use vaccine chatbot for the intervention group. Then, during the 1.5-month intervention, participants in the intervention group will be informed that the chatbot is available for use at their convenience, with coordinators sending the chatbot link every ten days to remind them to use. Conversely, the control group will not use the chatbot, without additional intervention during the trial, but will gain access after the trial ends.

At the end of the 1.5-month intervention, all participants from both intervention and control groups will be invited to complete a questionary survey. Three months after the intervention begins, influenza vaccination status of children and their parents will be collected from the vaccination registration system of local CDCs.

Difference in outcomes between the intervention and control groups will be assessed using t-tests and/or analysis of variance (ANOVA) for normally distributed continuous variables, and the Chi-square or Fisher's exact test will be used for categorical variables. When continuous variables do not meet normal distribution, the Wilcoxon rank-sum test will be employed. Multivariate regression models will be employed to evaluate the effectiveness of the chatbot intervention on the primary and secondary outcomes, adjusting for potential confounders. Given that participants in the intervention group will have varying frequencies and durations of using the chatbot, a dose-response relationship will be employed to evaluate the intervention effects by intervention intensity.

ELIGIBILITY:
Inclusion Criteria:

* Parents of the child visiting clinics.
* Children aged between 6 and 59 months.
* Children who have not received an influenza vaccine in both the current and previous flu seasons and have not yet made an appointment for an influenza vaccine.
* Children who have no contraindications to receiving an influenza vaccine.
* Provide informed consent and willing to participate throughout the study.

Exclusion Criteria:

* Children vaccinated or appointed for influenza vaccination or with any contraindication to influenza vaccine.
* Parents with mental disorders or visual/reading impairments, and unable to cooperate with and undergo the intervention activities.
* Unwilling to participate.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200 (Estimated)
Dates: Start 2024-10-26 (Estimated); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Influenza vaccination uptake for children | 1.5 months and three months
  whether the enrolled children receive an influenza vaccine. It will be measured in the survey at the end of the 1.5-month intervention, and be recorded from the vaccination registration system three months after the intervention begins.

SECONDARY OUTCOMES:
Influenza vaccination uptake for children's family members | 1.5 months and three months
  whether children's family members receive an influenza vaccine. It will be measured in the survey at the end of the 1.5-month intervention, and be recorded from the vaccination registration system three months after the intervention begins.
Influenza vaccination-specific consultation | 1.5 months
  whether parents consult health professionals about vaccinating their children with influenza vaccine during the 1.5-month intervention period, collected in the survey at the end of the 1.5-month intervention.
Influenza vaccine literacy | 1.5 months
  A series of ten questions about influenza vaccine knowledge and misinformation, collected in the survey at the end of the 1.5-month intervention. Total literacy score is calculated based on the number of questions answered correctly by the participants.
Influenza vaccine confidence | 1.5 months
  Vaccine Confidence Index, which evaluates parental perceptions of the vaccine's importance, effectiveness, and safety, collected in the survey at the end of the 1.5-month intervention.
Sustained vaccination intention | 1.5 months
  Whether parents intend to vaccinate their children against influenza in the next flu season, collected in the survey at the end of the 1.5-month intervention.

OTHER OUTCOMES:
Cost of chatbot intervention | 1.5 months
  The cost of designing vaccine chatbot and implementing chatbot intervention
Chatbot Usability | 1.5 months
  A series of questions assessing usability and feasibility, fairness and safety, user experience, and overall assessment of the chatbot.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyuan Hou, PhD, Principal Investigator — School of Public Health，Fudan University
Locations (1):
- Hangzhou Center for Disease Control and Prevention, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after de-identification (text, tables, figures, and appendices), will be shared upon reasonable requests. A written data-sharing request for meta-analysis should be submitted by email with a methodologically sound proposal. Proposals should be directed to zyhou@fudan.edu.cn; to gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol
Time Frame: Beginning 12 months and ending 36 months following article publication
Access Criteria: Researchers who provide a methodologically sound proposal for meta analysis. Proposals should be directed to zyhou@fudan.edu.cn; to gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Xianming C, Wu L, Chunyan Z, et al. Study of coverage of influenza and pneumonia vaccinations in children and influencing factors in two areas, China. Chinese Journal of Epidemiology. 2023;44(11):1731-1737.
- [Background] Nekrasova E, Stockwell MS, Localio R, Shults J, Wynn C, Shone LP, Berrigan L, Kolff C, Griffith M, Johnson A, Torres A, Opel DJ, Fiks AG. Vaccine hesitancy and influenza beliefs among parents of children requiring a second dose of influenza vaccine in a season: An American Academy of Pediatrics (AAP) Pediatric Research in Office Settings (PROS) study. Hum Vaccin Immunother. 2020 May 3;16(5):1070-1077. doi: 10.1080/21645515.2019.1707006. Epub 2020 Feb 4. PMID 32017643
- [Background] Szilagyi PG, Albertin CS, Saville AW, Valderrama R, Breck A, Helmkamp L, Zhou X, Vangala S, Dickinson LM, Tseng CH, Campbell JD, Whittington MD, Roth H, Rand CM, Humiston SG, Hoefer D, Kempe A. Effect of State Immunization Information System Based Reminder/Recall for Influenza Vaccinations: A Randomized Trial of Autodialer, Text, and Mailed Messages. J Pediatr. 2020 Jun;221:123-131.e4. doi: 10.1016/j.jpeds.2020.02.020. PMID 32446470
- [Background] Williams SE, Adams LE, Sommer EC. Improving Vaccination for Young Children (IVY): A Stepped-Wedge Cluster Randomized Trial. Acad Pediatr. 2021 Sep-Oct;21(7):1151-1160. doi: 10.1016/j.acap.2021.06.001. Epub 2021 Jun 10. PMID 34118498
- [Background] Lerner C, Albertin C, Casillas A, Duru OK, Ong MK, Vangala S, Humiston S, Evans S, Sloyan M, Fox CR, Bogard JE, Friedman S, Szilagyi PG. Patient Portal Reminders for Pediatric Influenza Vaccinations: A Randomized Clinical Trial. Pediatrics. 2021 Aug;148(2):e2020048413. doi: 10.1542/peds.2020-048413. PMID 34321338
- [Background] Stockwell MS, Shone LP, Nekrasova E, Wynn C, Torres A, Griffith M, Shults J, Unger R, Ware LA, Kolff C, Harris D, Berrigan L, Montague H, Localio AR, Fiks AG. Text Message Reminders for the Second Dose of Influenza Vaccine for Children: An RCT. Pediatrics. 2022 Sep 1;150(3):e2022056967. doi: 10.1542/peds.2022-056967. PMID 35965283
- [Background] Howell-Jones R, Gold N, Bowen S, Bunten A, Tan K, Saei A, Jones S, MacDonald P, Watson R, Bennett KF, Chadborn T. Can uptake of childhood influenza immunisation through schools and GP practices be increased through behaviourally-informed invitation letters and reminders: two pragmatic randomized controlled trials. BMC Public Health. 2023 Jan 20;23(1):143. doi: 10.1186/s12889-022-14439-4. PMID 36670376
- [Background] Szilagyi PG, Casillas A, Duru OK, Ong MK, Vangala S, Tseng CH, Albertin C, Humiston SG, Ross MK, Friedman SR, Evans S, Sloyan M, Bogard JE, Fox CR, Lerner C. Evaluation of behavioral economic strategies to raise influenza vaccination rates across a health system: Results from a randomized clinical trial. Prev Med. 2023 May;170:107474. doi: 10.1016/j.ypmed.2023.107474. Epub 2023 Mar 2. PMID 36870572
- [Background] Tuckerman J, Harper K, Sullivan TR, Cuthbert AR, Fereday J, Couper J, Smith N, Tai A, Kelly A, Couper R, Friswell M, Flood L, Blyth CC, Danchin M, Marshall HS. Short Message Service Reminder Nudge for Parents and Influenza Vaccination Uptake in Children and Adolescents With Special Risk Medical Conditions: The Flutext-4U Randomized Clinical Trial. JAMA Pediatr. 2023 Apr 1;177(4):337-344. doi: 10.1001/jamapediatrics.2022.6145. PMID 36806893
- [Background] Szilagyi PG, Duru OK, Casillas A, Ong MK, Vangala S, Tseng CH, Albertin C, Humiston SG, Clark E, Ross MK, Evans SA, Sloyan M, Fox CR, Lerner C. Text vs Patient Portal Messaging to Improve Influenza Vaccination Coverage: A Health System-Wide Randomized Clinical Trial. JAMA Intern Med. 2024 May 1;184(5):519-527. doi: 10.1001/jamainternmed.2024.0001. PMID 38497955